CLINICAL TRIAL: NCT02076100
Title: A Multiple Dose Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of MK-8408 in Subjects With Hepatitis C Infection
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of Ruzasvir (MK-8408) in Participants With Hepatitis C Infection (MK-8408-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8408-003; 2013-005094-41 (EudraCT Number); MK-8408-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I GT3 Participants (Experimental): Participants receive Ruzasvir capsules, orally, starting at a dose of 60 mg once per day (QD) x 5 days with doses increasing or decreasing as clinically indicated.
  Interventions: Drug: Ruzasvir
- Part II GT1a Participants (Experimental): Participants receive Ruzasvir capsules, orally, starting at a dose of 60 mg once per day (QD) x 5 days with doses increasing or decreasing as clinically indicated.
  Interventions: Drug: Ruzasvir
- Part III GT2b Participants (Experimental): Participants receive Ruzasvir capsules, orally, starting at a dose of 60 mg once per day (QD) x 5 days with doses increasing or decreasing as clinically indicated.
  Interventions: Drug: Ruzasvir

INTERVENTIONS:
Drug: Ruzasvir — Ruzasvir capsules, orally, starting at a dose of 60 mg once per day (QD) x 5 days with doses increasing or decreasing as clinically indicated.
  Other Names: MK-8408

SUMMARY:
This is a 3-part study of Ruzasvir (MK-8408) for participants with hepatitis C infection. Successive participants will be enrolled as dose levels are evaluated to find the maximum safe and well tolerated dose of Ruzasvir. Part I will be for participants with hepatitis C virus (HCV) genotype 3 (GT3) and will run first: Part II will be for participants with HCV genotype 1a (GT1a), and Part III will be for participants with HCV genotype 2b (GT2b). Parts II and III may run concurrently. The primary study hypothesis is that a safe and tolerable dose of Ruzasvir that reduces viral load will be found to support further clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >=18 to<=37 kg/m^2
* In general good health, except for HCV infection
* Clinical diagnosis of chronic HCV infection exclusively GT3 (Panels A-D) or exclusively GT1a (Panels E-F), or exclusively GT2b (Panels G-H).
* Must agree to follow the smoking restrictions defined by the CRU
* Must agree to use an acceptable method of contraception during the study and for 90 days after the last dose of ruzasvir

Exclusion Criteria:

* Clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormalities or diseases
* History of clinically significant hepatic disease, Gilbert's disease or biliary tract disease
* History of cancer (malignancy) with the exception of adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix, or successfully-treated malignancies ≥10 years prior to screening
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Positive for hepatitis B or human immunodeficiency virus (HIV)
* Major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to screening
* Participated in another investigational trial within 4 weeks prior to the screening visit
* QTc interval >=470 msec (for males) or >= 480 msec (for females)
* Unable to refrain from or anticipates use of any medication (prescription and/or non-prescription) or herbal remedies beginning approximately 2 weeks prior to first study drug dose, throughout the trial until the post-trial visit
* Consumes >2 glasses of alcoholic beverages per day
* Regular user (including "recreational use") of any illicit drugs or history of drug (including alcohol) abuse within approximately 12 months
* Evidence or history of chronic hepatitis not caused by HCV
* Previous treatment with other HCV NS5A inhibitors such as MK-8742, daclatasvir, or MK-8325
* Treatment with other HCV therapies such as the HCV protease
* Evidence of advanced or decompensated liver disease; evidence of bridging fibrosis or higher grade fibrosis (Metavir score >=3)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2015-11-15 (Actual); Study Completion 2015-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males or females of non-child bearing potential, with verified Hepatitis C virus (HCV) infection with genotype (GT) GT1a, GT2b or GT3 between the ages of 18 and 65 years (inclusive) were enrolled in this trial. In the GT1a group, one participant was later determined to be GT1b.
Groups:
- Ruzasvir 10 mg - GT3: GT3 participants were administered 10 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 30 mg - GT3: GT3 participants were administered 30 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 60 mg - GT3: GT3 participants were administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 120 mg - GT3: GT3 participants were administered 120 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 10 mg - GT2b: GT2b participants were administered 10 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 60 mg - GT2b: GT2b participants were administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 60 mg - GT1a: GT1a participants were administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days. One participant was later determined to be GT1b.
Period: Overall Study
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a
Started | 3 | 3 | 3 | 3 | 3 | 3 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (6.5) | 36.0 (3.5) | 38.0 (10.4) | 40.7 (13.6) | 56.3 (2.1) | 54.0 (6.2) | 48.5 (6.2) | 45.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Male | 2 | 3 | 3 | 3 | 2 | 2 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum log10 HCV Ribonucleic Acid (RNA) Change From Baseline
Description: Blood was collected at baseline and on Days 1, 2, 3, 4 and 5 to determine HCV RNA levels. Least squares means (LSM) and confidence intervals (CI) were obtained from an analysis of variance (ANOVA) model with maximum log10 HCV RNA change from baseline as response and a fixed effect for treatment. The primary hypothesis was that the mean change from baseline would be a reduction of ≥3 log10. A positive change from baseline indicates a reduction from baseline in log10 HCV RNA.
Time Frame: Baseline and up to Day 5
Population: Participants who complied with the protocol sufficiently to ensure that generated data would exhibit the effects of treatment, according to the underlying scientific model. Compliance covers considerations such as exposure to treatment, availability of measurements and absence of major protocol violations.
Measure: Least Squares Mean (90% Confidence Interval); unit: log10 IU/mL
Groups:
- Ruzasvir 60 mg - GT1a: GT1a participants were administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days.
- Ruzasvir 60 mg - GT1b: A GT1b participant was administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days.
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a | Ruzasvir 60 mg - GT1b
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1
log10 IU/mL | 2.84 [1.94 to 3.74] | 3.03 [2.13 to 3.94] | 3.36 [2.46 to 4.26] | 1.81 [0.90 to 2.71] | 3.82 [3.15 to 4.50] | 3.62 [2.95 to 4.30] | 3.63 [2.46 to 4.81] | 3.82 [NA to NA] — Data reflect n=1 and therefore 90% CI was not calculable.

2. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 61 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Ruzasvir 60 mg - GT3: Participants with GT3 were administered 60 mg Ruzasvir in capsule form, orally, once per day for 5 days.
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 4
Participants | 0 | 0 | 2 | 1 | 2 | 2 | 2

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due To An AE
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 5 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Ruzasvir 10 mg - GT3: Participants with GT3 were administered 10 mg Ruzasvir in capsule form, orally, once per day for 5 days.
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 61 days
Description: The population analyzed is all participants who received at least one dose of the investigational drug.
Arm/Group | Ruzasvir 10 mg - GT3 | Ruzasvir 30 mg - GT3 | Ruzasvir 60 mg - GT3 | Ruzasvir 120 mg - GT3 | Ruzasvir 10 mg - GT2b | Ruzasvir 60 mg - GT2b | Ruzasvir 60 mg - GT1a
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/3 | 1/3 | 2/3 | 2/3 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruzasvir 10 mg - GT3 (N=3) | Ruzasvir 30 mg - GT3 (N=3) | Ruzasvir 60 mg - GT3 (N=3) | Ruzasvir 120 mg - GT3 (N=3) | Ruzasvir 10 mg - GT2b (N=3) | Ruzasvir 60 mg - GT2b (N=3) | Ruzasvir 60 mg - GT1a (N=4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.